CLINICAL TRIAL: NCT00667758
Title: Antagonist to Gonadotropin-Releasing Hormone in Rheumatoid Arthritis (AGRA): A Double-blind, Randomized, Placebo Controlled Trial
Brief Title: Gonadotropin-Releasing Hormone (GnRH)-Antagonist Therapy in Rheumatoid Arthritis
Acronym: AGRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Betanien Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Anita Kass, Dr Anita Kåss, Betanien Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1/05; 2007/2/0174 (Other Grant/Funding Number: Norwegian Foundation for Health and Rehabilitation)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — cetrorelix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cetrorelix
  Interventions: Drug: Cetrorelix
- 2 (Placebo Comparator): NaCl solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cetrorelix — 3-5 mg s.c. on days 1-5
  Arms: 1
Drug: Placebo — 3-5 ml NaCl s.c. on days 1-5
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety and efficacy of gonadotropin-releasing hormone (GnRH) antagonist therapy versus placebo in patients with moderate to severe rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 years and above
* Moderate to severe disease activity
* Negative pregnancy test for women of childbearing potential
* Use of reliable method of contraception (non-hormonal) by sexually active female patients

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients taking biologic therapy or prednisolone >7.5mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in Disease Activity Score (DAS28CRP) in cetrorelix group versus placebo group | From baseline to day 5

SECONDARY OUTCOMES:
Change in DAS28 (CRP/ESR) | From baseline to day 2/5 /10/15
Change in anti-CCP level | From baseline to day 2/5/10/15
Change in cytokine level | From baseline to day 2/5/10/15
Change in ACR core set measures | From baseline to day 2/5/10/15
Proportion of patients with ACR 20/50/70/90 and EULAR good/moderate/none responders | Baseilne to day 2/5/10/15
Adverse events | Baseline up to day 15
  Number of patients with adverse events (and serious adverse events) up to day 15 in each group
Proportion of patients with DAS28low disease activity/remission | Baseline to day 2/5/10/15
Change in HAQ scores | From baseline to day 5/10/15
Correlation between percent changes in hormones, disease activity and biomarkers | By day 2, 5, 10 and 15
  This endpoint is not directly related to clinical efficacy. Hormones include LH, FSH, oestradiol, testosterone,and cortisol. Biomarkers include immunologic markers, bone markers and cardiovascular markers. This secondary endpoint was sent to authorities during the study before unblinding.

CONTACTS AND LOCATIONS:
Overall Officials: Kåss, Principal Investigator — University of Oslo
Locations (1):
- Deaprtment of Rheumatology, Betanien Hospital, Skien, Norway

REFERENCES:
- [Derived] Kass A, Hollan I, Fagerland MW, Gulseth HC, Torjesen PA, Forre OT. Rapid Anti-Inflammatory Effects of Gonadotropin-Releasing Hormone Antagonism in Rheumatoid Arthritis Patients with High Gonadotropin Levels in the AGRA Trial. PLoS One. 2015 Oct 13;10(10):e0139439. doi: 10.1371/journal.pone.0139439. eCollection 2015. PMID 26460564